CLINICAL TRIAL: NCT05389761
Title: Evaluation of the Efficacy of Fibromyalgia Treatment With Enzyme DAO (Diamine-oxidase)
Brief Title: Fibromyalgia Treatment With Enzyme DAO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centros de Investigación de Nutrición y Salud (Other)
Collaborators: AB Biotek (Industry)
Responsible Party: Principal Investigator, Ismael San Mauro Martin, Principal Investigator, Centros de Investigación de Nutrición y Salud
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2021/124-NUT-HRI
Record Dates: First submitted 2022-05-09; First posted 2022-05-25 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Diamine Oxidase; Supplementation; Genetics; Treatment
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enzyme DAO administration (Experimental): DAO enzyme supplementation for 6 months
  Interventions: Dietary Supplement: fibroDAO®
- Placebo administration (Placebo Comparator): Placebo supplementation for 6 months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: fibroDAO® — One DAO enzyme capsule is taken with water 20 minutes before each meal, 3 times a day. DAO enzyme capsules contains 0.3 mg DAO enzyme divided into 2 white/beige tablets (each gastro-resistant tablet contains 0.15 mg DAO enzyme) and 80 mg magnesium divided into 2 lilac tablets (each immediate-release tablet contains 40 mg of Mg).
  Arms: Enzyme DAO administration
Dietary Supplement: Placebo — One placebo capsule is taken with water 20 minutes before each meal, 3 times a day. Placebo capsules consist of microcrystalline cellulose and gelatin capsules with the same shape, size and colour as the DAO enzyme.
  Arms: Placebo administration

SUMMARY:
Fibromyalgia is a complex and common chronic pain disorder that affects 12 million Europeans. Fibromyalgia causes persistent widespread pain in muscles, tendons, ligaments, and joints, as well as widespread tenderness to touch and the presence of extreme fatigue and weakness.

Histamine is a molecule derived from an essential amino acid, histidine. It is stored in mast cells and basophils and is excreted through the intestine, being degraded as it passes through the intestinal mucosa by the enzyme Diamine Oxidase (DAO), which is found in this area. If there is any alteration in its metabolism and normal concentrations of histamine in the blood (50-70 mg/l) are not maintained, the free circulation of this amine in high concentrations triggers undesired effects, such as migraine, fibromyalgia, asthenia and atopy.

DAO deficiency is an alteration in the metabolism of dietary histamine that occurs when there is little activity of the DAO enzyme. The low activity of the enzyme causes that a concentration considered normal of histamine from food cannot be metabolized and a transepithelial penetration of exogenous histamine occurs. In this way, histamine passes into the bloodstream, increasing its plasma concentration and once located freely in the blood, it is distributed throughout different parts of the body, producing adverse effects.

One of the factors that causes DAO deficiency is genetics. The genetic sequence of DAO is found in a fragment located on chromosome 7 (7q34-q36) of the human genome. There are 85 single nucleotide variants (SNPs) located and identified in the human DAO gene (AOC1). Seven of these SNPs produce amino acid substitution, being candidates to cause alterations in the metabolic capacity of the enzyme.

Since histamine accumulation can trigger fibromyalgia, and the enzyme DAO has been shown to degrade histamine, oral supplementation with DAO food supplements, prepared from pig kidney, is suggested as a treatment for fibromyalgia.

The objective of this study is to analyze whether DAO enzyme supplementation reduces the characteristic symptoms of fibromyalgia. In addition, the prevalence of DAO deficiency in women with fibromyalgia will be identified by genetic analysis of DAO deficiency from a saliva sample. It will also be evaluated if patients require a lower intake of analgesics after supplementation with the enzyme DAO.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age between 30 and 59 years (included)
* Diagnosis of fibromyalgia
* Must sign an informed consent
* Able to follow-up at 2 and 6 months

Exclusion Criteria:

* Pregnant or possibly pregnant
* Patients with change of pharmacological treatment in the last 3 months
* Patients with DAO enzyme treatment
* Patients diagnosed with other severe diseases (i.e. cancer, cardiovascular disease, autoimmune disease or metabolic disease)
* Patients with multiple chemical sensitivity

Ages: 30 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
Patient status, progress and outcomes | Baseline, 2 months and 6 months
  Change from baseline in fibromyalgia status on the Fibromyalgia Impact Questionnaire (FIQ). The FIQ has10 items. Each item has a maximum possible score of 10. The maximum possible score is 100. A higher score indicates a greater impact of the syndrome.
Sleep quality | Baseline, 2 months and 6 months
  Change from baseline in sleep quality on the Pittsburgh Sleep Quality Index (PSQI). The PSQI contains 19 questions scored from 0 (no difficulty) to 3 (severe difficulty). The overall score is from 0 to 21. Higher scores indicate poorer sleep quality.
Pain experience | Baseline, 2 months and 6 months
  Change from baseline in pain on the Pain Catastrophizing Scale (PCS). The PCS contains 13 items that are rated on 5-point Likert scales, from 0 (not at all) to 4 (all the time). The minimum total score is 0 and the maximum is 52. A higher score indicates a higher level of catastrophizing.
Extent and severity of eczema | Baseline, 2 months and 6 months
  Change from baseline in eczema on the SCORing Atopic Dermatitis (SCORAD). The extension can be scored from 0 to 100, intensity from 0 to 18, and subjective symptoms from 0 to 20. The final score is achieved using the formula A / 5 + 7B / 2 + C.
Impact of headache | Baseline, 2 months and 6 months
  Change from baseline in headache on the Headache Impact Test-6 (HIT-6). HIT-6 has six questions, each with five response categories: never = 6, rarely = 8, sometimes = 10, very often = 11, and always = 13. The total score is obtained by adding the responses to the six items. Scores ≥ 60 indicate severe life impact, 56-59 substantial life impact, 50-55 some life impact, and ≤ 49 minimal or no life impact.

SECONDARY OUTCOMES:
Prevalence of DAO deficiency | Baseline
  Genetic analysis of DAO deficiency
Analgesic intake | Baseline, 2 months and 6 months
  Changes in analgesics intake. An ad-hoc questionnaire is used, where patients are asked to indicate the analgesics they take.

CONTACTS AND LOCATIONS:
Overall Officials: Ismael San Mauro Martin, PhD, Principal Investigator — Centros de Investigación de Nutrición y Salud
Locations (1):
- Hospital Ruber Internacional, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okutan G, Ruiz Casares E, Perucho Alcalde T, Sanchez Nino GM, Penades BF, Terren Lora A, Torrente Estringana L, Lopez Oliva S, San Mauro Martin I. Prevalence of Genetic Diamine Oxidase (DAO) Deficiency in Female Patients with Fibromyalgia in Spain. Biomedicines. 2023 Feb 22;11(3):660. doi: 10.3390/biomedicines11030660. PMID 36979637